CLINICAL TRIAL: NCT04984889
Title: An Open-Label, Single-Dose, Phase 1/2 Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Human Protein C (TAK-662) for the Treatment of Congenital Protein C Deficiency in Japanese Subjects Followed by an Extension Part
Brief Title: A Study of TAK-662 for Japanese Patients With Congenital Protein C Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-662-1501; U1111-1267-4412 (Other: WHO); jRCT2031210209 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-07-29; First posted 2021-08-02 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Congenital Protein C Deficiency
MeSH Terms: interventions — Protein C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAK-662 80 IU/kg (Experimental): TAK-662 80 international unit (IU)/kg, single intravenous infusion over 15 minutes on Day 1. In the extension part, dose of TAK-662 will be modified per participants. TAK-662 is Protein C Concentrate, which is a lyophilized, sterile concentrate of human protein C.
  Interventions: Drug: TAK-662

INTERVENTIONS:
Drug: TAK-662 — Lyophilized, sterile concentrate of human protein C
  Other Names: Protein C Concentrate

SUMMARY:
Pharmacokinetic Part:

This study is for Japanese participants with congenital protein C deficiency. The main aim of this study is to check how much TAK-662 stays in their blood over time. This will help the study sponsor (Takeda) to work out the best dose to give patients in the future.

Participants will receive 1 single infusion of TAK-662.

They will stay at the clinic until 3 days after the infusion. Then, participants will return to their clinic 7 days after the infusion to check side effects from the study treatment.

Extension Part:

Participants who will complete the PK part will be given an opportunity to continue TAK-662 administration as 3 different treatment options (on-demand therapy, short-term prophylaxis, and long-term prophylaxis) in the Extension part, until the commercial protein C concentrate is available at each study site or study termination.

ELIGIBILITY:
Inclusion Criteria:

PK Part:

1. Male and female participants with Japanese nationality.
2. A diagnosis of congenital protein C deficiency (homozygous or compound heterozygous).
3. Asymptomatic participant.
4. Oral anticoagulants allowed to be received.

Extension part:

1. Participants who participated in the PK part of this study (TAK-662-1501).
2. Participant who are; a. Diagnosed with PF, CISN/WISN, and/or other acute thromboembolic episode for on-demand treatment only; b. Requiring treatment with TAK-662 for short-term prophylaxis for surgical procedures; c. Requiring treatment with TAK-662 for long-term prophylaxis.

Exclusion Criteria:

PK Part:

1. Current or recurrent disease that could affect the action, or disposition of the investigational product (IP), or clinical or laboratory assessments.
2. A body weight less than 8 kg.
3. Serious liver dysfunction, judged by the investigator.
4. Any thrombosis within 2 weeks prior to administration of the IP.
5. Other investigational product than TAK-662 received within 60 days prior to the administration of the IP.
6. Current or relevant history of physical or psychiatric illness, or any medical disorder that may require treatment or make the participant unlikely to fully complete the study, or any condition that presents undue risk from the IP or procedures.
7. Current use of any medication (including over-the-counter, herbal, or homeopathic preparations) that could affect (improve or worsen) the condition being studied, or could affect the action or disposition of the IP, or clinical or laboratory assessment.
8. Known or suspected intolerance or hypersensitivity to the IP, closely-related compounds, or any of the stated ingredients.
9. Known history of alcohol or other substance abuse within the last year.
10. Within 30 days prior to the first dose of IP, a participant has been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this sponsored study.

Extension Part:

1. New serious medical conditions which could affect participant's safety or treatment were observed during participation in the PK part of this study (TAK-662-1501).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- Japan (4):
  - Nara Medical University Hospital, Kashihara, Nara
  - Chiba Children's Hospital, Chiba
  - Chiba University Hospital, Chiba
  - Saitama Prefectural Children's Medical Center, Saitama

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be reidentified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61081c16beb21d002a92609a

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 4 centers in Japan from 7 September 2021 to 31 October 2024.
Pre-assignment Details: A total of 5 Japanese participants were enrolled in this 2-part study to receive TAK-662 in Pharmacokinetic (PK) part (Part 1) followed by 3 treatment options in the Extension part (Part 2) (on-demand, short-term, or long-term prophylaxis). As per planned analysis, the Extension Part data was collected, analyzed and reported as per On-demand and Short-term Prophylaxis treatments and per dose level wise data was not collected in this study.
Groups:
- PK Part: TAK-662: Participants received a single 80 international unit per kilogram (IU/kg) dose of TAK-662, intravenous infusion on Day 1 in PK part.
- Extension Part, On-demand Treatment (TAK-662): Participants with purpura fulminans (PF), coumarin-induced skin necrosis/warfarin-induced skin necrosis (CISN/WISN), and/or other acute thromboembolic episode received a single dose of TAK-662 (100-120 IU/kg), followed by three subsequent infusions, every 6 hours at a dose of 60-80 IU/kg, and followed by subsequent infusions (45-60 IU/kg) continued every 6 or 12 hours until resolution of all non-necrotic lesions and/or stabilization of thrombi. Treatment could be terminated when an acute episode improved.
- Extension Part, Short-term Prophylaxis Treatment (TAK-662): Participants who required short-term prophylaxis of acute thrombotic episodes during surgery received TAK-662 at a dose of 100-120 IU/kg, intravenous infusion once daily, until anticoagulation therapy was successfully switched to TAK-662 prior to surgery. Fifteen minutes prior to surgery, a dose of 60-80 IU/kg was administered and continued once every 6 hours for the first 24 hours after surgery began. The frequency of infusions was reduced to 3 times daily between 24 and 48 hours, and twice daily after 48 hours at the same dose (45-60 IU/kg). Treatment with TAK-662 continued twice daily until anticoagulation therapy was initiated (if applicable) and the investigator determined that adequate level of the anticoagulation was achieved.
- Extension Part, Long-term Prophylaxis Treatment (TAK-662): Participants who required long-term prophylaxis were planned to receive TAK-662 at a dose of 45-60 IU/kg, intravenous infusion, twice daily. The dose was to be adjusted by referring to the latest protein C activity at the investigator's discretion. No participants received TAK-662 for long-term prophylaxis during the study.
Period: PK Part: Up to 7 Days
Arm/Group | PK Part: TAK-662 | Extension Part, On-demand Treatment (TAK-662) | Extension Part, Short-term Prophylaxis Treatment (TAK-662) | Extension Part, Long-term Prophylaxis Treatment (TAK-662)
Started | 5 | 0 | 0 | 0
Completed | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Extension Part: Up to 35 Months
Arm/Group | PK Part: TAK-662 | Extension Part, On-demand Treatment (TAK-662) | Extension Part, Short-term Prophylaxis Treatment (TAK-662) | Extension Part, Long-term Prophylaxis Treatment (TAK-662)
Started | 0 | 4 (Participants who completed PK Part and were eligible, received on-demand treatment in Extension Part.) | 1 (Participants who completed PK Part and were eligible, received short-term prophylaxis treatment in Extension Part.) | 0 (Participants who completed the PK part and were eligible to receive long-term prophylactic treatment in the extension part. However, no participant received the dose of TAK-662 for long-term prophylaxis.)
Completed | 0 | 4 | 1 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants in the study who took at least 1 dose of TAK-662.
Groups:
- PK Part: TAK-662: Participants received a single 80 IU/kg dose of TAK-662, intravenous infusion on Day 1 in PK part.
Arm/Group | PK Part: TAK-662
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 5

OUTCOME MEASURES:

1. Primary Outcome: PK Part: Protein C Activity Level of TAK-662
Description: Protein C is a vitamin K-dependent plasma protein and is an important component of the coagulation system. Protein C activity level was measured by chromogenic assays. Protein C activity level of TAK-662 was reported.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 12, 24, and 36 hours post-infusion
Population: The PK population included all study participants who took at least 1 dose of TAK-662 and had enough number of quantifiable blood levels for TAK-662 collected post-dose without important protocol deviations (PDs)/violations or events thought to substantially affect the PK.
Measure: Mean (Standard Deviation); unit: international unit per milliliter(IU/ml)
Arm/Group | PK Part: TAK-662
Number analyzed (Participants) | 5
international unit per milliliter(IU/ml)
  Pre-infusion | 0.000 (0.000)
  0.5 hour | 1.746 (0.557)
  1 hour | 1.616 (0.523)
  2 hours | 1.458 (0.519)
  4 hours | 1.168 (0.441)
  8 hours | 0.844 (0.295)
  12 hours | 0.632 (0.257)
  24 hours | 0.304 (0.150)
  36 hours | 0.148 (0.095)

2. Primary Outcome: PK Part: Terminal Phase Elimination Half-life (t1/2) of TAK-662
Description: t1/2 of TAK-662 was reported.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 12, 24, and 36 hours post-infusion
Population: The PK population included all study participants who took at least 1 dose of TAK-662 and had enough number of quantifiable blood levels for TAK-662 collected post-dose without important PDs/violations or events thought to substantially affect the PK.
Measure: Median (Full Range); unit: hour
Arm/Group | PK Part: TAK-662
Number analyzed (Participants) | 5
hour | 11.6 [7.68 to 13.0]

3. Primary Outcome: PK Part: Incremental Recovery (IR) of TAK-662
Description: IR of TAK-662 was reported measured in terms of international unit per milliliter/ international unit per kilogram (IU/mL)/(IU/kg).
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 12, 24, and 36 hours post-infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (IU/mL)/(IU/kg)
Arm/Group | PK Part: TAK-662
Number analyzed (Participants) | 5
(IU/mL)/(IU/kg) | 0.02063 (0.006588)

4. Primary Outcome: PK Part: Percentage of In-vivo Recovery (IVR) of TAK-662
Description: IVR corrected for plasma was determined using the formula: IVR (percentage [%])= (Maximum observed plasma concentration (Cmax) [IU/mL] - Concentration (C) pre-infusion [IU/mL]) * Plasma volume pre-infusion (PV) milliliter (mL)/ Dose (international unit [IU])*100 where Cmax was the observed Cmax value before baseline correction. IVR of TAK-662 measured in terms of percentage was reported.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 12, 24, and 36 hours post-infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of IVR
Arm/Group | PK Part: TAK-662
Number analyzed (Participants) | 5
percentage of IVR | 95.71 (31.22)

5. Primary Outcome: PK Part: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of TAK-662
Description: AUClast of TAK-662 was reported measured in terms of international unit*hour per milliliter (IU*h/ml).
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 12, 24, and 36 hours post-infusion
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*h/ml
Arm/Group | PK Part: TAK-662
Number analyzed (Participants) | 5
IU*h/ml | 19.24 (47.0)

6. Primary Outcome: PK Part: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-infinity) of TAK-662
Description: AUC0-infinity of TAK-662 was reported.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 12, 24, and 36 hours post-infusion
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU*h/ml
Arm/Group | PK Part: TAK-662
Number analyzed (Participants) | 5
IU*h/ml | 21.88 (47.1)

7. Primary Outcome: PK Part: Maximum Observed Plasma Concentration (Cmax) of TAK-662
Description: Cmax of TAK-662 was reported.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 12, 24, and 36 hours post-infusion
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/ml
Arm/Group | PK Part: TAK-662
Number analyzed (Participants) | 5
IU/ml | 1.679 (31.7)

8. Primary Outcome: PK Part: Time to Reach the Maximum Plasma Concentration (Tmax) of TAK-662
Description: Tmax of TAK-662 was reported.
Time Frame: Pre-infusion, 0.5, 1, 2, 4, 8, 12, 24, and 36 hours post-infusion
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | PK Part: TAK-662
Number analyzed (Participants) | 5
hour | 0.53 [0.43 to 0.60]

9. Secondary Outcome: PK and Extension Parts: Number of Participants With Treatment-Related Adverse Experiences (AEs)
Description: A treatment-related AE was defined as an adverse event that followed a reasonable temporal sequence from administration of a drug (including the course after withdrawal of the drug), or for which possible involvement of the drug was not able to be ruled out, although factors other than the drug, such as underlying diseases, complications, concomitant medications and concurrent treatments, might also be responsible. Number of participants with treatment-related AEs as assessed by the Investigator were reported.
Time Frame: PK Part: From the start of study drug administration up to Day 7; Extension Part: From the first dose of study drug administration in the Extension Part up to 35 months
Population: The safety population included all enrolled participants in the study who took at least 1 dose of TAK-662.
Measure: Count of Participants; unit: Participants
Groups:
- Extension Part, On-demand Treatment (TAK-662): Participants with PF, CISN/WISN, and/or other acute thromboembolic episode received a single dose of TAK-662 (100-120 IU/kg), followed by three subsequent infusions, every 6 hours at a dose of 60-80 IU/kg, and followed by subsequent infusions (45-60 IU/kg) continued every 6 or 12 hours until resolution of all non-necrotic lesions and/or stabilization of thrombi. Treatment could be terminated when an acute episode improved.
Arm/Group | PK Part: TAK-662 | Extension Part, On-demand Treatment (TAK-662) | Extension Part, Short-term Prophylaxis Treatment (TAK-662) | Extension Part, Long-term Prophylaxis Treatment (TAK-662)
Number analyzed (Participants) | 5 | 4 | 1 | 0
Participants | 1 | 0 | 0 | 0

10. Secondary Outcome: Extension Part: Number of Episode Rated as Effective, Effective With Complications, or Not Effective on Efficacy Rating Scale During On-Demand Treatment
Description: The treatment of episodes of PF, CISN/ WISN, and/or other vascular thromboembolic events were rated as "effective", "effective with complications", or "not effective" according to the efficacy rating scale, as judged by investigators on the basis of following criteria, Effective: stabilization and regression of skin lesions/stabilization of thrombi; Effective with complications: treatment was effective but caused an adverse drug reaction that interfered with the regimen (resulted in change of dose or frequency of dosing) or forcing discontinuation of treatment or introducing pathogenic viral infection; Not effective: all other cases.
Time Frame: Extension Part: From the first dose of TAK-662 on-demand treatment in the Extension Part up to 35 months
Population: Efficacy Analysis Set in On-Demand Treatment included all participants who took at least 1 dose of TAK-662 on-demand in the extension part.
Measure: Number; unit: treatment episodes
Units Other Than Participants: Total Number of Episodes
Arm/Group | Extension Part, On-demand Treatment (TAK-662)
Number analyzed (Participants) | 4
Number analyzed (Total Number of Episodes) | 19
treatment episodes
  Effective | 19
  Effective With Complications | 0
  Not Effective | 0

11. Secondary Outcome: Extension Part: Percentage of Surgical Episodes During Short-Term Prophylaxis That is Free of Presentations of PF or Thromboembolic Complications
Description: Percentage of surgical episodes for which TAK-662 was utilized as short-term prophylaxis that is free of presentations of PF or thromboembolic complications was reported.
Time Frame: Extension Part: From the first dose of TAK-662 short-term prophylaxis treatment in the Extension Part up to 35 months
Population: Efficacy Analysis Set in Short-term Prophylaxis included all participants who took at least 1 dose of TAK-662 during short-term prophylaxis in the extension part.
Measure: Number (95% Confidence Interval); unit: percentage of episode
Units Other Than Participants: Total Number of Surgical Episodes
Arm/Group | Extension Part, Short-term Prophylaxis Treatment (TAK-662)
Number analyzed (Participants) | 1
Number analyzed (Total Number of Surgical Episodes) | 1
percentage of episode | 100.0 [2.50 to 100.00]

12. Secondary Outcome: Extension Part: Number of Episodes of PF and/or Thrombotic Episodes During Long-Term Prophylaxis
Description: Number of episodes of PF and/or thrombotic episodes during long-term prophylaxis was planned to be reported.
Time Frame: Extension Part: From the first dose of TAK-662 long-term prophylaxis treatment in the Extension Part up to 35 months
Population: Efficacy Analysis Set in Long-term Prophylaxis included all study participants who took at least 1 dose of TAK-662 during long-term prophylaxis in the extension part. The "Overall Number of Participants Analyzed" is zero because no participants received TAK-662 for long-term prophylaxis; therefore, no data was collected and reported.
Arm/Group | Extension Part, Long-term Prophylaxis Treatment (TAK-662)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: PK Part: From start of study drug administration up to Day 7; Extension part: From first dose of study drug administration in Extension Part up to up to 35 months
Description: No participant received TAK-662 for long-term prophylaxis and therefore, no safety data could be collected and reported for 'Extension Part, Long-term Prophylaxis treatment (TAK-662) arm.
Arm/Group | PK Part: TAK-662 | Extension Part, On-demand Treatment (TAK-662) | Extension Part, Short-term Prophylaxis Treatment (TAK-662) | Extension Part, Long-term Prophylaxis Treatment (TAK-662)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 2/5 | 3/4 | 0/1 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PK Part: TAK-662 (N=5) | Extension Part, On-demand Treatment (TAK-662) (N=4) | Extension Part, Short-term Prophylaxis Treatment (TAK-662) (N=1) | Extension Part, Long-term Prophylaxis Treatment (TAK-662) (N=0)
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT04984889/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT04984889/SAP_001.pdf